CLINICAL TRIAL: NCT06564844
Title: A Phase III, Randomised, Open-label, Global Study of Adjuvant Datopotamab Deruxtecan (Dato-DXd) in Combination With Rilvegostomig or Rilvegostomig Monotherapy Versus Standard of Care, Following Complete Tumour Resection, in Participants With Stage I Adenocarcinoma Non-small Cell Lung Cancer Who Are ctDNA-positive or Have High-risk Pathological Features (TROPION-Lung12)
Brief Title: A Phase III, Randomised Study of Adjuvant Dato-DXd in Combination With Rilvegostomig or Rilvegostomig Monotherapy Versus Standard of Care, Following Complete Tumour Resection, in Participants With Stage I Adenocarcinoma NSCLC Who Are ctDNA-positive or Have High-risk Pathological Features
Acronym: TROPION-Lung12
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D926TC00001; 2024-512195-35-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-08-07; First posted 2024-08-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; NSCLC; Adenocarcinoma; Stage I; Datopotamab Deruxtecan; Dato-DXd; Adjuvant Treatment; Rilvegostomig; Standard of Care; Pemetrexed; Carboplatin; Cisplatin; Vinorelbine; Etoposide; UFT; ctDNA-positive; High-risk Pathological Features
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — Carboplatin; Cisplatin; Etoposide; Pemetrexed; Vinorelbine

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 2:1:2 ratio to one of the following groups: Arm 1 - Dato-DXd in combination with rilvegostomig, Arm 2 - rilvegostomig monotherapy or Arm 3 - SoC (either observation only or investigator's choice of chemotherapy (ICC)).
Who Masked: Outcomes Assessor
Masking Description: Open-label, sponsor-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dato-DXd + rilvegostomig (Experimental): Participants in the Dato-DXd in combination with rilvegostomig group will receive Dato-DXd and rilvegostomig as intravenous (IV) infusion every 3 weeks (Q3W).
  Interventions: Drug: Datopotamab Deruxtecan; Drug: Rilvegostomig
- Rilvegostomig (Experimental): Participants in the rilvegostomig monotherapy group will receive rilvegostomig as intravenous (IV) infusion every 3 weeks (Q3W).
  Interventions: Drug: Rilvegostomig
- Standard of Care (SoC) (Active Comparator): Patients in SoC group will undergo observation or will receive Investigator's Choice of Chemotherapy (ICC).
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Drug: Pemetrexed; Drug: Vinorelbine; Drug: UFT

INTERVENTIONS:
Drug: Datopotamab Deruxtecan — Datopotamab Deruxtecan IV (intravenous)
  Other Names: Dato-DXd, DS-1062a
  Arms: Dato-DXd + rilvegostomig
Drug: Rilvegostomig — Rilvegostomig IV (intravenous)
  Other Names: AZD2936
  Arms: Dato-DXd + rilvegostomig; Rilvegostomig
Drug: Carboplatin — Carboplatin IV (intravenous), Active Comparator
  Arms: Standard of Care (SoC)
Drug: Cisplatin — Cisplatin IV (intravenous), Active Comparator
  Arms: Standard of Care (SoC)
Drug: Etoposide — Etoposide IV (intravenous), Active Comparator
  Arms: Standard of Care (SoC)
Drug: Pemetrexed — Pemetrexed IV (intravenous), Active Comparator
  Arms: Standard of Care (SoC)
Drug: Vinorelbine — Vinorelbine IV (intravenous), Active Comparator
  Arms: Standard of Care (SoC)
Drug: UFT — UFT Oral route of administration, Active Comparator
  Arms: Standard of Care (SoC)

SUMMARY:
This is a Phase III, randomised, open-label, multicentre, global study assessing the efficacy and safety of adjuvant Dato-DXd in combination with rilvegostomig compared with SoC, after complete surgical resection (R0) in participants with Stage I adenocarcinoma NSCLC who are ctDNA-positive, as determined by the Sponsor-designated ctDNA assay, or have at least one high-risk pathological feature.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the efficacy and safety of adjuvant Dato-DXd in combination with rilvegostomig relative to SoC, after complete surgical resection (R0) in participants with Stage I adenocarcinoma NSCLC who are ctDNA-positive, as determined by the Sponsor-designated ctDNA assay, or have at least one high-risk pathological feature.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented treatment-naive Stage I (T < 4 cm, AJCC 8th ed) adenocarcinoma NSCLC
2. Complete surgical resection (R0) of the primary NSCLC
3. Unequivocal no evidence of disease at post-surgical
4. Pre-surgical ctDNA-positive result (Stage IA or IB) OR presence of at least one high-risk pathological feature (visceral pleural invasion (VPI), lymphovascular invasion (LVI), high-grade histology) (Stage IB only)
5. ECOG of 0 or 1, life expectancy of > 6 months and complete recovery after surgery
6. Adequate bone marrow reserve and organ function

Exclusion Criteria:

1. Sensitizing EGFR mutation and/or ALK alteration
2. History of non-infectious ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
3. Significant pulmonary function compromise
4. History of another primary malignancy within 3 years (with exceptions)
5. Any evidence of severe or uncontrolled systemic diseases, including but not limited to bleeding diseases, active infection and cardiac disease
6. Active or prior documented autoimmune or inflammatory disorders (with exceptions)
7. Active infection with tuberculosis, hepatitis B or C virus, hepatitis A, or known HIV infection that is not well controlled
8. History of active primary immunodeficiency
9. Clinically significant corneal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) using BICR in participants with Stage I adenocarcinoma NSCLC who are ctDNA-positive or having at least one high-risk pathological feature treated with adjuvant Dato-DXd in combination with rilvegostomig relative to SoC | From date of randomisation up to approximately 10 years.
  The analysis will include all randomised participants as randomised. All events will be included, regardless of whether the participant withdraws from randomised therapy or receives another anti-cancer therapy.
  The measure of interest is the HR of DFS.
  Descriptive analyses of Dato-DXd in combination with rilvegostomig versus rilvegostomig monotherapy and rilvegostomig monotherapy versus SoC will be performed to assess contribution of components.

SECONDARY OUTCOMES:
Overall Survival (OS) in participants with Stage I adenocarcinoma NSCLC who are ctDNA-positive or having at least one high-risk pathological feature treated with adjuvant Dato-DXd in combination with rilvegostomig relative to SoC | From date of randomisation up to approximately 10 years.
  The analysis will include all randomised participants as randomised. All deaths will be included, regardless of whether the participant withdraws from therapy or receives another anti-cancer therapy.
  The measure of interest is the HR of OS.
  Descriptive analyses of Dato-DXd in combination with rilvegostomig versus rilvegostomig monotherapy and rilvegostomig monotherapy versus SoC will be performed to assess contribution of components.
Participant-reported physical function in participants with Stage I adenocarcinoma NSCLC who are ctDNA-positive or having at least one high-risk pathological feature treated with adjuvant Dato-DXd in combination with rilvegostomig relative to SoC | Measured at weeks 12, 24 and 48.
  The analysis will include all randomised participants as randomised. The physical function will be measured by the PROMIS SF PF 8c. Data from PROMIS SF PF 8c will capture participants' perceived ability to perform specific activities from daily life and will be scored on a 5-point rating scale.
  The measure of interest will be the between treatment group difference in adjusted mean in physical function scores.
  Descriptive analyses of Dato-DXd in combination with rilvegostomig versus rilvegostomig monotherapy and rilvegostomig monotherapy versus SoC will be performed to assess contribution of components.
Participant-reported GHS/QoL in participants with Stage I adenocarcinoma NSCLC who are ctDNA-positive or having at least one high-risk pathological feature treated with adjuvant Dato-DXd in combination with rilvegostomig relative to SoC | Measured at weeks 12, 24 and 48.
  The analysis will include all randomised participants as randomised. The GHS/QoL scores will be measured by the GHS/QoL scale from EORTC IL172.
  The measure of interest will be the between treatment group difference in adjusted mean in GHS/QoL scores.
  Descriptive analyses of Dato-DXd in combination with rilvegostomig versus rilvegostomig monotherapy and rilvegostomig monotherapy versus SoC will be performed to assess contribution of components.
Pharmacokinetics (PK) | Up to 30 or 90 days post-last dose of study intervention.
  Concentration of Dato-DXd, total anti-TROP2 antibody, and MAAA-1181a (payload deruxtecan) in plasma or serum.
Pharmacokinetics (PK) | Up to 30 or 90 days post-last dose of study intervention.
  Concentration of rilvegostomig in plasma or serum.
Pharmacokinetics (PK) | Up to 30 or 90 days post-last dose of study intervention.
  PK parameters (peak and through concentrations).
Immunogenicity | Up to 30 or 90 days post-last dose of study intervention.
  Presence of ADAs for Dato-DXd and rilvegostomig (confirmatory results: titres and neutralising antibodies for confirmed positive samples).

CONTACTS AND LOCATIONS:
Overall Officials: David Jones, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center, New York, United States of America; Enriqueta Felip, MD, Principal Investigator — Vall d'Hebron Hospital, Barcelona, Spain
Locations (90):
- United States (37):
  - Research Site, Tucson, Arizona
  - Research Site, Duarte, California
  - Research Site, Glendale, California
  - Research Site, Los Angeles, California
  - Research Site, Lone Tree, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Zion, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Farmington Hills, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Billings, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, East Syracuse, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Edmonds, Washington
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Brazil (5):
  - Research Site, Barretos
  - Research Site, Brasília
  - Research Site, Florianópolis
  - Research Site, São Paulo
  - Research Site, Teresina
- Canada (5):
  - Research Site, Halifax, Nova Scotia
  - Research Site, Oshawa, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Research Site, Hong Kong, Hong Kong
- Japan (19):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Hiroshima
  - Research Site, Iwakuni-shi
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Wakayama
  - Research Site, Yokohama
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Bangkoknoi
  - Research Site, Banphaeo
  - Research Site, Dusit
  - Research Site, Hat Yai
  - Research Site, Muang
  - Research Site, Ratchathewi
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Mersin
- United Kingdom (3):
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Nottingham
- Vietnam (5):
  - Research Site, Da Nang
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
  For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool.
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home